CLINICAL TRIAL: NCT05628350
Title: Reducing Highly Processed Foods to Improve Vascular Health in Middle-Aged Adults
Brief Title: Highly Processed Foods and Vascular Health
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Virginia Polytechnic Institute and State University (Other)
Collaborators: Duke University (Other)
Responsible Party: Principal Investigator, Kevin Davy, Professor, Virginia Polytechnic Institute and State University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 22-819
Record Dates: First submitted 2022-11-16; First posted 2022-11-28 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Cardiovascular Diseases
Keywords: Middle age; Diet composition; Vascular function
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- No UPF (Ultra-processed foods) (Experimental): Following a 2-week eucaloric lead-in diet, participants will be provided and consume a diet without UPF (0% total energy) for 6 weeks.
  Interventions: Other: No UPF controlled diet
- High UPF (Experimental): Following a 2-week eucaloric lead-in diet, participants will be provided and consume a diet composed of 81% UPF for 6 weeks.
  Interventions: Other: High UPF controlled diet

INTERVENTIONS:
Other: No UPF controlled diet — Following a two-week eucaloric lead-in diet, participants will be provided and consume a diet without UPF (0% total energy) for 6 weeks. Diets will be eucaloric (50% carbohydrate, 35% fat, 15% protein) and matched for dietary soluble and insoluble fiber, added sugar, mono- and polyunsaturated fat, saturated fat, antioxidant nutrients, sodium, pre- and probiotics, and overall diet quality.
  Arms: No UPF (Ultra-processed foods)
Other: High UPF controlled diet — Following a two-week eucaloric lead-in diet, participants will be provided and consume a diet with high UPF intake (81% total energy) for 6 weeks. Diets will be eucaloric (50% carbohydrate, 35% fat, 15% protein) and matched for dietary soluble and insoluble fiber, added sugar, mono- and polyunsaturated fat, saturated fat, antioxidant nutrients, sodium, pre- and probiotics, and overall diet quality.
  Arms: High UPF

SUMMARY:
Age is the primary risk factor for cardiovascular disease (CVD) and age-related vascular dysfunction is considered the key process linking the two. Middle age is a particularly vulnerable period when risk factors exceed diagnostic thresholds and clinical expression of CVD first becomes evident. Ultra-processed foods (UPF) comprise almost 60% of total energy in the standard American diet. The results of observational studies suggest that UPF consumption increases CVD risk, independent of overall diet quality (i.e., saturated fat, sodium, sugar, and dietary fiber intake). The "industrialized microbiota" may link diet, particularly UPF, to increased inflammation and CVD in middle-aged adults. High intake of UPF increases the likelihood of an excess heart age >10 years and doubles the risk of subclinical coronary atherosclerosis in middle-aged adults. However, the impact of reducing UPF consumption on vascular function in middle-aged adults is unknown. The overall objective of this study is to establish proof-of-concept for an improvement in vascular function following reductions in UPF consumption in mid-life adults, in order to conduct a larger, more comprehensive and mechanistic trial in the future. In addition, changes in gut microbial composition and function, intestinal inflammation and permeability, serum endotoxin concentrations, and inflammatory cytokines as potential mechanisms by which UPF consumption influences vascular function will be investigated.

ELIGIBILITY:
Inclusion Criteria:

* Weight stable for previous 6 months (<2 kg change)
* Sedentary to recreationally active
* No plans to gain/lose weight or change physical activity level
* Willing to pick up food daily and consume foods provided for an 8-week period
* Verbal and written informed consent
* Approval by Medical Director
* Usual UPF intake +/-15% of US average of 60% total energy
* Estrogen or testosterone usage is acceptable, if on stable dose for >6 months
* Lipid-lowering medication usage is acceptable, if on a stable dose for >6 months

Exclusion Criteria:

* BMI >35 kg/m2
* Diabetes or diabetes medication
* Antibiotic, prebiotic or prebiotic use in prior 3 months
* Total Cholesterol >6.2 mmol/L; Triglycerides >4.5 mmol/L
* Blood pressure (BP) > 159/99 mmHg (Stable BP on antihypertensive medications is acceptable)
* Diagnosed inflammatory bowel disease
* Past or current heart diseases, stroke, respiratory disease, endocrine or metabolic disease, or hematological-oncological disease
* Vegetarian or vegan
* Pregnant or plans to become pregnant
* Food allergies or aversions
* 3 or fewer stools per week or regular laxative use
* Lipid-lowering medication usage <6 months

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2023-07-19 (Actual); Primary Completion 2024-12-18 (Actual); Study Completion 2025-09-30 (Actual)

PRIMARY OUTCOMES:
Change in brachial artery function from baseline to 6-weeks post no or high UPF diet | 30-minute measurement in the laboratory, 2 timepoints (baseline, 6 weeks post no or high UPF diet)
  Flow Mediated Dilation (FMD) of the brachial artery will be assessed using duplex ultrasonography (GE Logiq e) with a high-resolution linear array transducer. Reactive hyperemia will be produced by inflation of a pediatric BP cuff around the forearm for 5 minutes. Offline analysis of baseline and post-reactive hyperemic diameters and velocities will be performed using edge detection software (Vascular Analysis Tools, Medical Imaging Applications, Inc). Endothelium independent vasodilation (EID) will be assessed by measuring brachial arterial dilation for 10 minutes following administration of 0.4 mg of sublingual nitroglycerine. Both FMD and EID will be expressed as mm and % change from baseline diameter.

SECONDARY OUTCOMES:
Change in arterial stiffness (Carotid femoral pulse wave velocity) from baseline to 6-weeks post no or high UPF diet | 45-minute measurement in the laboratory, 2 timepoints (baseline, 6 weeks post no or high UPF diet)
  Carotid femoral (C-F) pulse wave velocity (PWV), the primary measure of arterial stiffness, will be measured. C-F waveforms will be obtained via tonometry (NIHem, Cardiovascular Engineering, Inc). Aortic PWV will be calculated from signal averaged waveforms using the ECG as the fiducial point, and body surface measurements.
Change in gut microbial composition from baseline to post 6-weeks no or high UPF diet | 3-day collection during free-living, 2 timepoints (baseline, 6 weeks post no or high UPF diet)
  Stool samples will be collected daily for 3 days before and during the final 3 days of the diet interventions. Samples will be collected daily and placed in sterile plastic containers, stored in personal freezers, and placed in coolers for transport. Upon return to the lab, they will be immediately frozen at -80°C until final processing and analysis.
Change in gut microbial function from baseline to post 6-weeks no or high UPF diet | 3-day collection during free-living, 2 timepoints (baseline, 6 weeks post no or high UPF diet)
  Stool samples will be collected daily for 3 days before and during the final 3 days of the diet interventions. Samples will be collected daily and placed in sterile plastic containers, stored in personal freezers, and placed in coolers for transport. Upon return to the lab, they will be immediately frozen at -80°C until final processing and analysis.
Change in intestinal inflammation from baseline to post 6-weeks no or high UPF diet | 3-day collection during free-living, 2 timepoints (baseline, 6 weeks post no or high UPF diet)
  Intestinal inflammation will be assessed using fecal calprotectin, lactoferrin, and lipocalin-2, measured using ELISA.
Change in intestinal permeability from baseline to post 6-weeks no or high UPF diet | 3-day collection during free-living, 2 timepoints (baseline, 6 weeks post no or high UPF diet)
  Intestinal permeability will be assessed using serum zonulin (Immunodiagnostik AG, Bensheim, Germany) concentrations, measured using ELISA.
Change in inflammatory cytokines from baseline to post 6-weeks no or high UPF diet | 5-minute blood collection in the laboratory, 2 timepoints (baseline, 6 weeks post no or high UPF diet)
  Inflammatory cytokines, including Tumor Necrosis Factor alpha, Interleukin 6, and Monocyte Chemoattractant Protein-1, will be measured using ELISA (American Diagnostica Inc).
Change in endotoxin from baseline to post 6-weeks no or high UPF diet | 5-minute blood collection in the laboratory, 2 timepoints (baseline, 6 weeks post no or high UPF diet)
  Serum endotoxin will be assessed using the PyroGene Recombinant Factor C endotoxin assay (Lonza, Basel, Switzerland).

OTHER OUTCOMES:
Change in insulin sensitivity from baseline to 6-weeks post no or high UPF diet | 2-hour test in laboratory, 2 timepoints (baseline, 6-weeks post no or high UPF diet)
  Insulin sensitivity assessed using a 2-hour oral glucose tolerance test (75g glucose load). Blood will be collected at baseline (fasting), and thereafter, at 30-minute intervals (5 total measurements in 2 hours).
Change in 24-hour glucose control (24-hour mean) from baseline to 6-weeks post no or high UPF diet | 6-day measurement during free-living, 2 timepoints (baseline, 6 weeks post no or high UPF diet)
  24-hour glucose control (24-hour mean glucose concentration) will be assessed using continuous glucose monitoring for a 6-day period.
Change in 24-hour glucose control (AUC) from baseline to 6-weeks post no or high UPF diet | 6-day measurement during free-living, 2 timepoints (baseline, 6 weeks post no or high UPF diet)
  24-hour glucose control (24-hour AUC) will be assessed using continuous glucose monitoring for a 6-day period.
Change in 24-hour glucose control (time in range) from baseline to 6-weeks post no or high UPF diet | 6-day measurement during free-living, 2 timepoints (baseline, 6 weeks post no or high UPF diet)
  24-hour glucose control (time in range) will be assessed using continuous glucose monitoring for a 6-day period.
Change in 24-hour glucose control (glycemic variability [GV]) from baseline to 6-weeks post no or high UPF diet | 6-day measurement during free-living, 2 timepoints (baseline, 6 weeks post no or high UPF diet)
  24-hour glucose control (GV) will be assessed using continuous glucose monitoring for a 6-day period.
Change in 24-hour glucose control (postprandial glucose) from baseline to 6-weeks post no or high UPF diet | 6-day measurement during free-living, 2 timepoints (baseline, 6 weeks post no or high UPF diet)
  Free-living postprandial glucose concentration will be assessed using continuous glucose monitoring for a 6-day period.

CONTACTS AND LOCATIONS:
Overall Officials: Kevin Davy, PhD, Principal Investigator — Virginia Polytechnic Institute and State University
Locations (1):
- Virginia Polytechnic and State University, Blacksburg, Virginia, United States

IPD SHARING:
Plan to Share IPD: No